CLINICAL TRIAL: NCT00524355
Title: Epidemiological Study to Assess the Symptoms and Patterns of Diagnosis and Treatment of the Gastroesophageal Reflux Disease
Brief Title: Epidemiological Study to Assess the Symptoms and Patterns of Diagnosis and Treatment of GERD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-GVN-NEX-2007/1; NIS-G84-GER-2007/2
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2009-07-17 (Estimated); Status verified 2009-07

CONDITIONS: GERD
Keywords: GERD; GIS; heartburn; NIS; PPI
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe the frequency, type and severity of the symptoms in patients visiting the GI or internal physicians, with symptoms consistent with gastroesophageal reflux disease (GERD)

ELIGIBILITY:
Inclusion Criteria:

* Patients from both sexes, aged 18 years or older
* Patients complaining of symptoms consistent with reflux disease

Exclusion Criteria:

* Patients with GI cancer and those where the only reason for the visit is renewing the prescription are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinics, private clinics and out-patient department at hospitals in cities and provinces of Viet Nam
Sampling Method: Probability Sample
Enrollment: 2717 (Actual)
Dates: Start 2007-03; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ta Long, MD, PhD, Study Chair — 108 Hospital, Hanoi; Do Van Dung, MD, PhD, Study Chair — Ho Chi Minh City Univ of Medicine and Pharmacist; Dao Van Long, MD, PhD, Principal Investigator — Ha Noi University of Medicine Hospital
Locations (2):
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City